CLINICAL TRIAL: NCT02373488
Title: The Effects of Connective Tissue Manipulation and Abdominal Massage in Patients With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceren Gürşen, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 14/480
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Constipation
Keywords: Constipation; connective tissue manipulation; abdominal massage; bowel movements; quality of life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Other): lifestyle advice
  Interventions: Other: lifestyle advice
- intervention-1 (Active Comparator): connective tissue manipulation
  Interventions: Other: lifestyle advice; Other: connective tissue manipulation
- intervention-2 (Active Comparator): abdominal massage
  Interventions: Other: lifestyle advice; Other: abdominal massage

INTERVENTIONS:
Other: lifestyle advice — lifestyle advices such as increasing fluid and fibre intake, improving physical activity level, and taking the ideal posture for defecation (squatting position) with a two-pages document.
Other: connective tissue manipulation — CTM wil be applied five days per week, a total of 20 sessions for 4 weeks. Each session lasted around 15-20 minutes. While patients are in a sitting position, starting from the lumbosacral region, lower thoracic, scapular, inter-scapular and cervical regions will be included in the treatment, respectively.
  Arms: intervention-1
Other: abdominal massage — Abdominal massage will be applied five days a week for four weeks. Each session will last around 15-20 minutes.
  Arms: intervention-2

SUMMARY:
The aim of this study is to investigate the effect of connective tissue manipulation and abdominal massage on severity of constipation and health related quality of life in patients with chronic constipation. According to literature, there are studies that investigate the effects of abdominal massage on bowel movements. But there is no randomized controlled trial, explore the short and long-term effects of different massage technics on chronic constipation. Hypothesis of this study is that connective tissue manipulation and abdominal massage improves symptoms of constipation and health related quality of life in patients suffering with constipation.

DETAILED DESCRIPTION:
Chronic constipation is not a disease but a symptom of a condition involving insufficient defecation and whose definition varies from person to person. Health professionals define constipation as 3 times or less per week defecation and the patients define it as the sensation of incomplete bowel evacuation, hard stool, straining, and difficulty in defecation. Chronic constipation is a common condition experienced by the general public, and it reduces the health related quality of life (HRQOL) by negatively affecting the physical, mental, and social well being of individuals. In a recent meta-analysis, the global prevalence rate of chronic constipation was reported to be 14%; it was also reported that its incidence rate is correlated with increasing age and low-income level, and it is more common among females.

Because the underlying pathophysiology of chronic constipation has not been clearly identified, its treatment has been difficult for both healthcare professionals and patients. Following the elimination of pathological and secondary causes, the treatment of chronic constipation is initiated by non-pharmacological treatment methods, such as lifestyle modifications (increased dietary fiber and water intake as well as increased physical activity), defecation training, and physiotherapy approaches. If lifestyle modification and conservative treatment methods do not help the patient, pharmacological treatment methods, such as osmotic laxatives, stimulant laxatives, stool softeners, lubricants, chloride channel activators, and serotonin agents, may be used. At the final stage, if the pharmacological treatment is not successful in patients with slow-transit constipation, surgical treatment options, such as segmental, subtotal, or total colectomy, are considered. Conservative treatment methods used in patients with chronic constipation may include abdominal massage, connective tissue manipulation (CTM), chiropractic treatment, electrical stimulation, anorectal biofeedback and exercise.

CTM, one of the conservative treatment methods for chronic constipation, generates local mechanical effects on mast cells in the connective tissue by short and long tractions and thus creates vasodilation by reducing the sympathetic activity. Subsequently, parasympathetic effect increases and the improvement in the circulation promotes healing process. But there is very little research that examine its effectiveness on constipation and bowel function. In the case report of Holey et al., it was reported that CTM was better than abdominal massage in improving symptoms of constipation. Also, another study revealed that combination of pelvic exercises and CTM played a role in healing bowel functions in women immediately after the post cesarean delivery.

Abdominal massage is another treatment approach using the management of chronic constipation. The benefits of physiotherapy in treatment of constipation include mechanical and neurological effects. Mechanical effects include accelerating colonic motility, improving colonic transit time, coordinating the muscles and increasing abdominal muscle tone. The neurological effect is to enhance the activity of the parasympathetic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be recruited if they were over 18 years of age and had a diagnosis of chronic constipation according to Rome III criteria. Rome III classification system is widely use and standardized symptom-based diagnostic criteria for functional gastrointestinal disorders, including chronic constipation. Rome III criteria include that having at least 2 of the following: 1) straining; 2) lumpy and hard stool; 3) sensation of incomplete evacuation; 4) sensation of anorectal obstruction/blockage; 5) need for manual maneuvers 6) fewer than three defecation during ≥ 25% defecations. Also, symptoms should begin at least six months prior the diagnosis and they should be seen intermittently or continuously for three months.

Exclusion Criteria:

* comorbid neurological, anatomical, or metabolic condition, pregnancy, mental problems preventing cooperation, history of colostomy surgery, history of gastrointestinal, spinal, or pelvic surgery except cholecystectomy, appendectomy, or hysterectomy, comorbid various colonic conditions (intestinal obstruction, peritonitis, bowel perforation, peptic ulcer, gastrointestinal bleeding, or acute inflammation of abdominal organs), history of intestinal cancer, existence of open sore or tumor at the massage region, and abdominal hernia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
severity of constipation | change from baseline severity of constipation at 4 weeks
  Constipation Severity Instrument (CSI) will be used to evaluate the severity of the constipation. CSI was designed to evaluate defecation frequency and consistency as well as the level of straining experienced by individuals during bowel movement. There are three subscales of CSI, obstructive defecation (OT), colonic inertia (CI), and pain. Higher scores of CSI indicate more severe constipation.

SECONDARY OUTCOMES:
Stool consistency | change from baseline stool consistency at 4 weeks
  The stool consistency will be evaluated using the Bristol Stool Scale (BSS), quick and useful indicator of the colonic transit time , a seven-point scale (from 1 to 7), type 1=separate hard lumps, like nuts; 2=sausage shaped but lumpy; 3=like a sausage or snake, but with cracks on its surface; 4=like a sausage or snake, smooth and soft; 5=soft blobs with clear cut edges; 6=ﬂuffy pieces with ragged edges, a mushy stool; 7=water, no solid pieces. While type 1 and 2 indicate hard stool, type 3,4 and 5 show looser (ideal) stool.
symptoms of constipation | change from baseline symptoms of constipation at 4 weeks
  In order to gather information regarding the participants' symptoms of constipation, they will be asked to complete a 7-day bowel diary during the treatment period. This diary includes items regarding the frequency of bowel movement, stool consistency, defecation time, feeling of incomplete evacuation, and changes in food and liquid consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Lamas K, Lindholm L, Stenlund H, Engstrom B, Jacobsson C. Effects of abdominal massage in management of constipation--a randomized controlled trial. Int J Nurs Stud. 2009 Jun;46(6):759-67. doi: 10.1016/j.ijnurstu.2009.01.007. Epub 2009 Feb 12. PMID 19217105
- [Background] Sinclair M. The use of abdominal massage to treat chronic constipation. J Bodyw Mov Ther. 2011 Oct;15(4):436-45. doi: 10.1016/j.jbmt.2010.07.007. Epub 2010 Aug 25. PMID 21943617
- [Background] Holey LA, Dixon J, Selfe J. An exploratory thermographic investigation of the effects of connective tissue massage on autonomic function. J Manipulative Physiol Ther. 2011 Sep;34(7):457-62. doi: 10.1016/j.jmpt.2011.05.012. Epub 2011 Jul 23. PMID 21875520
- [Background] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158